CLINICAL TRIAL: NCT00111475
Title: A Dose-finding Study Evaluating the Safety and Efficacy of AMG 531 in Thrombocytopenic Subjects With Immune Thrombocytopenic Purpura (ITP)
Brief Title: Evaluating the Safety and Efficacy of Romiplostim (AMG 531) in Thrombocytopenic Subjects With Immune Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20000137
Record Dates: First submitted 2005-05-20; First posted 2005-05-23 (Estimated); Results first posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2019-12

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: Immune Thrombocytopenic Purpura; Idiopathic Thrombocytopenic Purpura; Thrombocytopenic; Thrombocytopenia; ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia | interventions — romiplostim

STUDY DESIGN:
Intervention Model Description: Part A was a sequential cohort dose escalation study. Part B was a randomized, placebo-controlled parallel group study.
Who Masked: Participant, Investigator

ARMS (10):
- Part A: Romiplostim 0.2 µg/kg (Experimental): Participants received 0.2 µg/kg romiplostim subcutaneously on day 1 and day 15 or 22, depending on platelet counts.
  Interventions: Drug: Romiplostim
- Part A: Romiplostim 0.5 µg/kg (Experimental): Participants received 0.5 µg/kg romiplostim subcutaneously on day 1 and day 15 or 22, depending on platelet counts.
  Interventions: Drug: Romiplostim
- Part A: Romiplostim 1.0 µg/kg (Experimental): Participants received 1.0 µg/kg romiplostim subcutaneously on day 1 and on day 15 or 22 depending on platelet counts.
  Interventions: Drug: Romiplostim
- Part A: Romiplostim 3 µg/kg (Experimental): Participants received 3.0 µg/kg romiplostim subcutaneously on day 1 and day 15 or 22, depending on platelet counts.
  Interventions: Drug: Romiplostim
- Part A: Romiplostim 6 µg/kg (Experimental): Participants received 6.0 µg/kg romiplostim subcutaneously on day 1 and day 15 or 22, depending on platelet counts.
  Interventions: Drug: Romiplostim
- Part A: Romiplostim 10 µg/kg (Experimental): Participants received 10.0 µg/kg romiplostim subcutaneously on day 1 and day 15 or 22, depending on platelet counts.
  Interventions: Drug: Romiplostim
- Part B: Placebo (Placebo Comparator): Participants received placebo subcutaneously once a week for 6 weeks.
  Interventions: Drug: Placebo
- Part B: Romiplostim 1.0 µg/kg (Experimental): Participants received 1.0 µg/kg subcutaneously once a week for 6 weeks.
  Interventions: Drug: Romiplostim
- Part B: Romiplostim 3.0 µg/kg (Experimental): Participants received 3.0 µg/kg subcutaneously once a week for 6 weeks.
  Interventions: Drug: Romiplostim
- Part B: Romiplostim 6.0 µg/kg (Experimental): Participants received 6.0 µg/kg subcutaneously once a week for 6 weeks.
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim — Administered by subcutaneous injection
  Other Names: AMG 531; NPLATE
  Arms: Part A: Romiplostim 0.2 µg/kg; Part A: Romiplostim 0.5 µg/kg; Part A: Romiplostim 1.0 µg/kg; Part A: Romiplostim 10 µg/kg; Part A: Romiplostim 3 µg/kg; Part A: Romiplostim 6 µg/kg; Part B: Romiplostim 1.0 µg/kg; Part B: Romiplostim 3.0 µg/kg; Part B: Romiplostim 6.0 µg/kg
Drug: Placebo — Administered by subcutaneous injection
  Arms: Part B: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of romiplostim in thrombocytopenic patients with ITP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ITP according to American Society of Hematology (ASH) guidelines at least 3 months before enrollment
* Have completed at least 1 prior treatment for ITP
* Two (including day -2) of the 3 platelet counts taken during the screening and pre-treatment periods must have fulfilled the following:

  * less than 30 x 10^9/L for those subjects not receiving any ITP therapy,
  * less than 50 x 10^9/L for those subjects receiving any ITP therapy
* Eastern Cooperative Oncology Group performance status of 0 to 2
* Serum creatinine concentration ≤ 2 mg/dL (≤ 176.8 µmol/L)
* Adequate liver function, as evidenced by a serum bilirubin ≤ 1.5 times the laboratory normal range
* Hemoglobin greater than 10.0 g/dL
* Written informed consent

Exclusion Criteria:

* Considered a substantial risk for adverse outcomes because of a clinically important trend (as determined by the investigator) detected in the platelet counts during the screening period
* Any known history of bone marrow stem cell disorder
* Any active malignancy. If prior history of cancer other than basal cell carcinoma or cervical carcinoma in situ, no treatment or active disease within 5 years before randomization
* Documented diagnosis of arterial thrombosis (ie, stroke, transient ischemic attack, or myocardial infarction) in the previous year; history of venous thrombosis (ie, deep vein thrombosis, pulmonary embolism) and receiving anticoagulation therapy
* Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure [New York Heart Association (NYHA) greater than class II], uncontrolled hypertension [diastolic greater than 100 mmHg] or cardiac arrhythmia)
* Have 3 or more of the following predisposing factors for thromboembolic events: diabetes; smoker using oral contraceptives; hypercholesteremia (> 240 mg/dL); treatment for hypertension
* Known positive test for human immunodeficiency virus (HIV) infection or hepatitis C virus
* Received any treatment for ITP (except for a constant dose schedule of corticosteroids) within 4 weeks before the screening visit
* Received intravenous (IV) immunoglobulin (Ig) or WinRho within 2 weeks before the screening visit
* Received hematopoietic growth factors, including interleukin (IL)-11 (Neumega®) within 4 weeks before the screening visit
* Past or present participation in any study evaluating polyethylene glycol recombinant human magakaryopoiesis differentiating factor (PEG-rHuMGDF), recombinant human thrombopoietin (rHuTPO), or related platelet product
* Received any alkylating agents within 8 weeks before the screening visit or anticipated use during the time of the proposed study
* Received any monoclonal antibody (eg, rituximab) within 16 weeks before the screening visit or anticipated use during the time of the proposed study
* Less than 4 weeks since receipt of any therapeutic drug or device that is not FDA approved for any indication before the screening period
* Less than 2 months since major surgery (including laparoscopic splenectomy)
* Pregnant or breast feeding
* Subjects of reproductive potential who are not using adequate contraceptive precautions, in the judgment of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2002-07-01 (Actual); Primary Completion 2004-06-17 (Actual); Study Completion 2004-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Cines DB, Wasser J, Rodeghiero F, Chong BH, Steurer M, Provan D, Lyons R, Garcia-Chavez J, Carpenter N, Wang X, Eisen M. Safety and efficacy of romiplostim in splenectomized and nonsplenectomized patients with primary immune thrombocytopenia. Haematologica. 2017 Aug;102(8):1342-1351. doi: 10.3324/haematol.2016.161968. Epub 2017 Apr 14. PMID 28411254
- [Background] Bussel JB, Kuter DJ, George JN, McMillan R, Aledort LM, Conklin GT, Lichtin AE, Lyons RM, Nieva J, Wasser JS, Wiznitzer I, Kelly R, Chen CF, Nichol JL. AMG 531, a thrombopoiesis-stimulating protein, for chronic ITP. N Engl J Med. 2006 Oct 19;355(16):1672-81. doi: 10.1056/NEJMoa054626. PMID 17050891
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_46_AMP-2_20000137.pdf
- See also: FDA-approved Drug Labeling — http://www.nplate.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of 2 parts. Part A (conducted from July 1, 2002 to October 13, 2003) was an open-label, dose-escalation trial with sequential cohorts of participants.
  Part B (conducted from October 6, 2003 to June 17, 2004) was a double-blind, placebo-controlled, parallel design study.
Pre-assignment Details: In Part A participants were sequentially assigned to escalating dose cohorts. In Part B, participants were randomized to each dose cohort; within each cohort 2 of 10 participants were randomly assigned to receive placebo. The 6.0 µg/kg dose cohort was discontinued in protocol amendment 4.
Groups:
- Part A: Romiplostim 0.2 µg/kg: Participants received 0.2 µg/kg romiplostim on day 1 and day 15 or 22, depending on platelet counts
- Part A: Romiplostim 0.5 µg/kg: Participants received 0.5 µg/kg romiplostim on day 1 and day 15 or 22, depending on platelet counts.
- Part A: Romiplostim 1.0 µg/kg: Participants received 1.0 µg/kg romiplostim on day 1 and on day 15 or 22 depending on platelet counts.
- Part A: Romiplostim 3 µg/kg: Participants received 3.0 µg/kg romiplostim on day 1 and day 15 or 22, depending on platelet counts.
- Part A: Romiplostim 6 µg/kg: Participants received 6.0 µg/kg romiplostim on day 1 and day 15 or 22, depending on platelet counts.
- Part A: Romiplostim 10 µg/kg: Participants received 10.0 µg/kg romiplostim on day 1 and day 15 or 22, depending on platelet counts.
- Part B: Placebo: Participants received placebo by subcutaneous injection once a week for 6 weeks.
- Part B: Romiplostim 1.0 µg/kg: Participants received 1.0 µg/kg romiplostim by subcutaneous injection once a week for 6 weeks.
- Part B: Romiplostim 3.0 µg/kg: Participants received 3.0 µg/kg romiplostim by subcutaneous injection once a week for 6 weeks.
- Part B: Romiplostim 6.0 µg/kg: Participants received 6.0 µg/kg romiplostim by subcutaneous injection once a week for 6 weeks.
Period: Overall Study
Arm/Group | Part A: Romiplostim 0.2 µg/kg | Part A: Romiplostim 0.5 µg/kg | Part A: Romiplostim 1.0 µg/kg | Part A: Romiplostim 3 µg/kg | Part A: Romiplostim 6 µg/kg | Part A: Romiplostim 10 µg/kg | Part B: Placebo | Part B: Romiplostim 1.0 µg/kg | Part B: Romiplostim 3.0 µg/kg | Part B: Romiplostim 6.0 µg/kg
Started | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 8 | 8 | 1
Completed | 4 | 4 | 4 | 4 | 4 | 3 | 4 | 8 | 8 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Romiplostim 0.2 µg/kg | Part A: Romiplostim 0.5 µg/kg | Part A: Romiplostim 1.0 µg/kg | Part A: Romiplostim 3 µg/kg | Part A: Romiplostim 6 µg/kg | Part A: Romiplostim 10 µg/kg | Part B: Placebo | Part B: Romiplostim 1.0 µg/kg | Part B: Romiplostim 3.0 µg/kg | Part B: Romiplostim 6.0 µg/kg | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 8 | 8 | 1 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Part A and Part B were analyzed separately; no overall total was calculated.
  years
    Part A: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 24
    Part A | 43.5 (15.0) | 42.8 (11.1) | 42.5 (10.7) | 44.8 (18.2) | 41.3 (14.7) | 47.5 (14.5) |  |  |  |  | 43.7 (12.8)
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 8 | 8 | 1 | 21
    Part B |  |  |  |  |  |  | 53.0 (10.6) | 43.0 (15.0) | 47.4 (16.6) | 42.0 (NA) — N=1 | 14.3 (49.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4 | 4 | 3 | 2 | 3 | 6 | 5 | 1 | 32
  Male | 1 | 3 | 0 | 0 | 1 | 2 | 1 | 2 | 3 | 0 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 4 | 4 | 4 | 3 | 3 | 3 | 5 | 5 | 1 | 36
  Black | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3
  Hispanic | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 6
Plateleet Count [Mean (Standard Deviation); unit: 1 × 10⁹ cells/L] — Population: Part A and Part B were analyzed separately; no overall total was calculated.
  1 × 10⁹ cells/L
    Part A: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 24
    Part A | 10.7 (2.70) | 14.5 (12.5) | 9.06 (4.19) | 13.4 (6.81) | 12.6 (9.00) | 18.4 (10.1) |  |  |  |  | 13.1 (7.93)
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 8 | 8 | 1 | 21
    Part B |  |  |  |  |  |  | 28.4 (17.7) | 16.9 (7.86) | 14.0 (6.20) | 15.0 (NA) — N=1 | 17.9 (10.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: From first dose of study drug through 8 weeks (Part A) or 6 weeks (Part B) after last dose of study drug; 78 days
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Romiplostim 0.2 µg/kg | Part A: Romiplostim 0.5 µg/kg | Part A: Romiplostim 1.0 µg/kg | Part A: Romiplostim 3 µg/kg | Part A: Romiplostim 6 µg/kg | Part A: Romiplostim 10 µg/kg | Part B: Placebo | Part B: Romiplostim 1.0 µg/kg | Part B: Romiplostim 3.0 µg/kg | Part B: Romiplostim 6.0 µg/kg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 8 | 8 | 1
Participants
  Any adverse event | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 8 | 8 | 1
  Serious adverse events | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0
  Treatment-related adverse events | 0 | 0 | 3 | 0 | 1 | 1 | 1 | 2 | 4 | 0
  Treatment-related serious adverse events | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Discontinuations due to adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Anti-romiplostim or Anti-endogenous Thrombopoietin Neutralizing Antibodies
Description: The development of antibodies to romiplostim or to endogenous thrombopoietin (eTPO) was assessed using a neutralizing bioassay. Participants positive for neutralizing antibodies at any of the assessments during the study are reported.
Time Frame: Assessed on day 29 (Part A only), day 43 (Part B only), and day 78
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Romiplostim 0.2 µg/kg | Part A: Romiplostim 0.5 µg/kg | Part A: Romiplostim 1.0 µg/kg | Part A: Romiplostim 3 µg/kg | Part A: Romiplostim 6 µg/kg | Part A: Romiplostim 10 µg/kg | Part B: Placebo | Part B: Romiplostim 1.0 µg/kg | Part B: Romiplostim 3.0 µg/kg | Part B: Romiplostim 6.0 µg/kg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 8 | 8 | 1
Participants
  Anti-romiplostim neutralizing antibodies | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anti-eTPO neutralizing antibodies | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants Who Achieved Targeted Therapeutic Platelet Level in Part A
Description: Targeted therapeutic platelet level was defined as a doubling of baseline platelet counts and between 50 to 450 x 10⁹ cells/L.
  Platelet count data after the use of rescue medication were not included; participants with no platelet count data were considered non-responders.
Time Frame: After first dose (day 1 to day 15 or 22) and after second dose (day 15 or 22 to day 78)
Population: Participants enrolled in Part A who received each dose of romiplostim.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Romiplostim 0.2 µg/kg | Part A: Romiplostim 0.5 µg/kg | Part A: Romiplostim 1.0 µg/kg | Part A: Romiplostim 3 µg/kg | Part A: Romiplostim 6 µg/kg | Part A: Romiplostim 10 µg/kg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
Participants
  After first dose | 1 | 0 | 0 | 1 | 1 | 1
  After second dose: number analyzed (Participants) | 3 | 4 | 4 | 4 | 3 | 2
  After second dose | 1 | 0 | 0 | 2 | 1 | 1
  After both doses: number analyzed (Participants) | 3 | 4 | 4 | 4 | 3 | 2
  After both doses | 1 | 0 | 0 | 1 | 1 | 1

4. Secondary Outcome: Number of Participants With an Increase in Platelet Count of ≥ 20 x 10⁹ Cells/L Over Baseline in Part A
Description: Platelet count data after the use of rescue medication were not included; participants with no platelet count data were considered non-responders.
Time Frame: After first dose (day 1 to day 15 or 22), and after second dose (day 15 or 22 to day 78)
Population: Participants enrolled in Part A who received each dose of romiplostim
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Romiplostim 0.2 µg/kg | Part A: Romiplostim 0.5 µg/kg | Part A: Romiplostim 1.0 µg/kg | Part A: Romiplostim 3 µg/kg | Part A: Romiplostim 6 µg/kg | Part A: Romiplostim 10 µg/kg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
Participants
  After first dose | 1 | 1 | 1 | 2 | 2 | 3
  After second dose: number analyzed (Participants) | 3 | 4 | 4 | 4 | 3 | 2
  After second dose | 1 | 0 | 0 | 3 | 1 | 1
  After both doses: number analyzed (Participants) | 3 | 4 | 4 | 4 | 3 | 2
  After both doses | 1 | 0 | 0 | 2 | 1 | 1

5. Secondary Outcome: Number of Participants With a Peak Platelet Count ≥ 100 x 10⁹ Cells/L in Part A
Description: as for outcome 4
Time Frame: After first dose (day 1 to day 15 or 22) and after second dose (day 15 or 22 to day 78)
Population: Participants enrolled in Part A who received each dose of romiplostim
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Romiplostim 0.2 µg/kg | Part A: Romiplostim 0.5 µg/kg | Part A: Romiplostim 1.0 µg/kg | Part A: Romiplostim 3 µg/kg | Part A: Romiplostim 6 µg/kg | Part A: Romiplostim 10 µg/kg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
Participants
  After first dose | 1 | 0 | 0 | 1 | 2 | 3
  After second dose: number analyzed (Participants) | 3 | 4 | 4 | 4 | 3 | 2
  After second dose | 0 | 0 | 0 | 2 | 1 | 1
  After both doses: number analyzed (Participants) | 3 | 4 | 4 | 4 | 3 | 2
  After both doses | 0 | 0 | 0 | 1 | 1 | 1

6. Secondary Outcome: Number of Participants With a Peak Platelet Count of > 450 x 10⁹ Cells/L in Part A
Description: as for outcome 4
Time Frame: After first dose (day 1 to day 15 or 22) and after second dose (day 15 or 22 to day 78)
Population: Participants enrolled in Part A who received each dose of romiplostim
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Romiplostim 0.2 µg/kg | Part A: Romiplostim 0.5 µg/kg | Part A: Romiplostim 1.0 µg/kg | Part A: Romiplostim 3 µg/kg | Part A: Romiplostim 6 µg/kg | Part A: Romiplostim 10 µg/kg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
Participants
  After first dose | 0 | 0 | 0 | 0 | 1 | 2
  After second dose: number analyzed (Participants) | 3 | 4 | 4 | 4 | 3 | 2
  After second dose | 0 | 0 | 0 | 0 | 0 | 0
  After both doses: number analyzed (Participants) | 3 | 4 | 4 | 4 | 3 | 2
  After both doses | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Peak Platelet Count After Each Dose in Part A
Description: Platelet count data after the use of rescue medication were not included.
Time Frame: After first dose (day 1 to day 15 or 22) and after second dose (day 15 or 22 to day 78)
Population: Participants enrolled in Part A who received each dose of romiplostim and with a platelet count of ≥ 50 × 10⁹ cells/L and a doubling of the baseline platelet count, in the absence of rescue medication.
Measure: Mean (Standard Deviation); unit: 1 × 10⁹ cells/L
Arm/Group | Part A: Romiplostim 0.2 µg/kg | Part A: Romiplostim 0.5 µg/kg | Part A: Romiplostim 1.0 µg/kg | Part A: Romiplostim 3 µg/kg | Part A: Romiplostim 6 µg/kg | Part A: Romiplostim 10 µg/kg
Number analyzed (Participants) | 1 | 0 | 0 | 2 | 2 | 3
1 × 10⁹ cells/L
  After first dose: number analyzed (Participants) | 1 | 0 | 0 | 1 | 2 | 3
  After first dose | 123.0 |  |  | 163.0 | 309.0 (202.2) | 746.3 (611.9)
  After second dose: number analyzed (Participants) | 1 | 0 | 0 | 2 | 1 | 1
  After second dose | 65.0 |  |  | 140.5 (29.0) | 244.0 | 259.0

8. Secondary Outcome: Change From Baseline in Peak Platelet Count After Each Dose in Part A
Description: Platelet count data after the use of rescue medication were not included.
Time Frame: Baseline and after first dose (day 1 to day 15 or 22) and after second dose (day 15 or 22 to day 78)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 1 × 10⁹ cells/L
Arm/Group | Part A: Romiplostim 0.2 µg/kg | Part A: Romiplostim 0.5 µg/kg | Part A: Romiplostim 1.0 µg/kg | Part A: Romiplostim 3 µg/kg | Part A: Romiplostim 6 µg/kg | Part A: Romiplostim 10 µg/kg
Number analyzed (Participants) | 1 | 0 | 0 | 2 | 2 | 3
1 × 10⁹ cells/L
  After first dose: number analyzed (Participants) | 1 | 0 | 0 | 1 | 2 | 3
  After first dose | 109.5 |  |  | 150.2 | 289.3 (208.2) | 725.5 (622.5)
  After second dose: number analyzed (Participants) | 1 | 0 | 0 | 2 | 1 | 1
  After second dose | 51.50 |  |  | 122.6 (21.78) | 220.0 | 231.7

9. Secondary Outcome: Time to Peak Platelet Count After Each Dose in Part A
Description: Platelet count data after the use of rescue medication were not included.
Time Frame: After first dose (day 1 to day 15 or 22) and after second dose (day 15 or 22 to day 78)
Population: as for outcome 7
Measure: Median (Full Range); unit: days
Arm/Group | Part A: Romiplostim 0.2 µg/kg | Part A: Romiplostim 0.5 µg/kg | Part A: Romiplostim 1.0 µg/kg | Part A: Romiplostim 3 µg/kg | Part A: Romiplostim 6 µg/kg | Part A: Romiplostim 10 µg/kg
Number analyzed (Participants) | 1 | 0 | 0 | 2 | 2 | 3
days
  After first dose: number analyzed (Participants) | 1 | 0 | 0 | 1 | 2 | 3
  After first dose | 10.0 [10 to 10] |  |  | 11.0 [11 to 11] | 9.5 [8 to 11] | 15.0 [12 to 15]
  After second dose: number analyzed (Participants) | 1 | 0 | 0 | 2 | 1 | 1
  After second dose | 10.0 [10 to 10] |  |  | 11.0 [9 to 13] | 10.0 [10 to 10] | 11.0 [11 to 11]

10. Secondary Outcome: Duration Within the Targeted Therapeutic Platelet Range In Part A
Description: Targeted therapeutic platelet level was defined as a platelet count that was double the baseline level and ≥ 50 and ≤ 450 × 10⁹ cells/L.
  Platelet count data after the use of rescue medication were not included.
Time Frame: After first dose (day 1 to day 15 or 22) and after second dose (day 15 or 22 to day 78)
Population: Participants enrolled in Part A who received each dose of romiplostim and with a platelet count ≥ 50 × 10⁹ cells/L and ≤ 450 × 10⁹ cells/L and a doubling of the baseline platelet count, in the absence of rescue medication.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Part A: Romiplostim 0.2 µg/kg | Part A: Romiplostim 0.5 µg/kg | Part A: Romiplostim 1.0 µg/kg | Part A: Romiplostim 3 µg/kg | Part A: Romiplostim 6 µg/kg | Part A: Romiplostim 10 µg/kg
Number analyzed (Participants) | 1 | 0 | 0 | 2 | 1 | 1
days
  After first dose: number analyzed (Participants) | 1 | 0 | 0 | 1 | 1 | 1
  After first dose | 5.0 |  |  | 8.0 | 11.0 | 10.0
  After second dose | 3.0 |  |  | 3.5 (2.1) | 11.0 | 9.0

11. Secondary Outcome: Percentage of Participants Who Achieved Targeted Therapeutic Platelet Level In Part B
Description: Targeted therapeutic platelet level was defined as a doubling of baseline platelet counts and within the range of greater than or equal to 50 x 10⁹ cells/L and less than or equal to 450 x 10⁹ cells/L.
  Platelet count data after use of rescue medication were not included in the analysis.
Time Frame: Day 1 to day 78
Population: Participants randomized in Part B who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Placebo | Part B: Romiplostim 1.0 µg/kg | Part B: Romiplostim 3.0 µg/kg | Part B: Romiplostim 6.0 µg/kg
Number analyzed (Participants) | 4 | 8 | 8 | 1
percentage of participants | 25 | 88 | 38 | 0

12. Secondary Outcome: Percentage of Participants With an Increase in Platelet Count of ≥ 20 x 10⁹ Cells/L Over Baseline in Part B
Description: Platelet count data after administration of rescue medication were not included in the analysis. Participants with no platelet count data were considered non-responders.
Time Frame: Day 1 to day 78
Population: Participants randomized in Part B who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Placebo | Part B: Romiplostim 1.0 µg/kg | Part B: Romiplostim 3.0 µg/kg | Part B: Romiplostim 6.0 µg/kg
Number analyzed (Participants) | 4 | 8 | 8 | 1
percentage of participants | 50 | 100 | 75 | 100

13. Secondary Outcome: Percentage of Participants With a Peak Platelet Count of ≥ 100 x 10⁹ Cells/L in Part B
Description: as for outcome 12
Time Frame: Day 1 to day 78
Population: Participants randomized in Part B who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Placebo | Part B: Romiplostim 1.0 µg/kg | Part B: Romiplostim 3.0 µg/kg | Part B: Romiplostim 6.0 µg/kg
Number analyzed (Participants) | 4 | 8 | 8 | 1
percentage of participants | 25 | 63 | 63 | 100

14. Secondary Outcome: Percentage of Participants With a Peak Platelet Count of > 450 x 10⁹ Cells/L in Part B
Description: as for outcome 12
Time Frame: Day 1 to day 78
Population: Participants randomized in Part B who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Placebo | Part B: Romiplostim 1.0 µg/kg | Part B: Romiplostim 3.0 µg/kg | Part B: Romiplostim 6.0 µg/kg
Number analyzed (Participants) | 4 | 8 | 8 | 1
percentage of participants | 0 | 0 | 25 | 100

15. Secondary Outcome: Percentage of Participants With a Peak Platelet Count of > 500 x 10⁹ Cells/L in Part B
Description: as for outcome 12
Time Frame: Day 1 to day 78
Population: Participants randomized in Part B who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Placebo | Part B: Romiplostim 1.0 µg/kg | Part B: Romiplostim 3.0 µg/kg | Part B: Romiplostim 6.0 µg/kg
Number analyzed (Participants) | 4 | 8 | 8 | 1
percentage of participants | 0 | 0 | 25 | 100

16. Secondary Outcome: Peak Platelet Count in Part B
Description: Platelet count data after administration of rescue medication were not included in the analysis.
Time Frame: Day 1 to day 78
Population: Participants randomized in Part B who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: 1 × 10⁹ cells/L
Arm/Group | Part B: Placebo | Part B: Romiplostim 1.0 µg/kg | Part B: Romiplostim 3.0 µg/kg | Part B: Romiplostim 6.0 µg/kg
Number analyzed (Participants) | 4 | 8 | 8 | 1
1 × 10⁹ cells/L | 80.8 (96.0) | 134.5 (90.2) | 240.9 (288.3) | 520.0

17. Secondary Outcome: Change From Baseline in Peak Platelet Count in Part B
Description: Platelet count data after administration of rescue medication were not included in the analysis.
Time Frame: Baseline and day 1 to day 78
Population: Participants randomized in Part B who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: 1 × 10⁹ cells/L
Arm/Group | Part B: Placebo | Part B: Romiplostim 1.0 µg/kg | Part B: Romiplostim 3.0 µg/kg | Part B: Romiplostim 6.0 µg/kg
Number analyzed (Participants) | 4 | 8 | 8 | 1
1 × 10⁹ cells/L | 52.4 (92.9) | 117.6 (88.3) | 226.9 (284.1) | 505.0

18. Secondary Outcome: Time to Peak Platelet Count in Part B
Description: Platelet count data after administration of rescue medication were not included in the analysis. Time to peak platelet count was analyzed using the Kaplan-Meier method.
Time Frame: Day 1 to day 78
Population: Participants randomized in Part B who received at least 1 dose of study drug.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Part B: Placebo | Part B: Romiplostim 1.0 µg/kg | Part B: Romiplostim 3.0 µg/kg | Part B: Romiplostim 6.0 µg/kg
Number analyzed (Participants) | 4 | 8 | 8 | 1
days | 63 [27.5 to 78] | 18 [11.5 to 35.5] | 19 [11 to 35.5] | 21 [21 to 21]

19. Secondary Outcome: Duration Within the Targeted Therapeutic Platelet Range in Part B
Description: Targeted therapeutic platelet level was defined as a doubling of baseline platelet counts and within the range of greater than or equal to 50 × 10⁹ cells/L and less than or equal to 450 × 10⁹ cells/L.
  Platelet count data after administration of rescue medication were not included in the analysis.
Time Frame: Day 1 to day 78
Population: Participants randomized in Part B who received at least 1 dose of study drug and achieved a targeted therapeutic platelet level.
Measure: Median (Full Range); unit: weeks
Arm/Group | Part B: Placebo | Part B: Romiplostim 1.0 µg/kg | Part B: Romiplostim 3.0 µg/kg | Part B: Romiplostim 6.0 µg/kg
Number analyzed (Participants) | 1 | 7 | 5 | 1
weeks | 6.0 [6 to 6] | 3.0 [1 to 7] | 5.0 [1 to 7] | 4.0 [4 to 4]

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 8 weeks (Part A) or 6 weeks (Part B) after last dose of study drug; 78 days.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Part A: Romiplostim 0.2 µg/kg | Part A: Romiplostim 0.5 µg/kg | Part A: Romiplostim 1.0 µg/kg | Part A: Romiplostim 3 µg/kg | Part A: Romiplostim 6 µg/kg | Part A: Romiplostim 10 µg/kg | Part B: Placebo | Part B: Romiplostim 1.0 µg/kg | Part B: Romiplostim 3.0 µg/kg | Part B: Romiplostim 6.0 µg/kg
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/4 | 0/4 | 0/4 | 0/4 | 1/4 | 2/4 | 0/8 | 1/8 | 0/1
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4 | 4/4 | 4/4 | 4/4 | 4/4 | 8/8 | 8/8 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Romiplostim 0.2 µg/kg (N=4) | Part A: Romiplostim 0.5 µg/kg (N=4) | Part A: Romiplostim 1.0 µg/kg (N=4) | Part A: Romiplostim 3 µg/kg (N=4) | Part A: Romiplostim 6 µg/kg (N=4) | Part A: Romiplostim 10 µg/kg (N=4) | Part B: Placebo (N=4) | Part B: Romiplostim 1.0 µg/kg (N=8) | Part B: Romiplostim 3.0 µg/kg (N=8) | Part B: Romiplostim 6.0 µg/kg (N=1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Romiplostim 0.2 µg/kg (N=4) | Part A: Romiplostim 0.5 µg/kg (N=4) | Part A: Romiplostim 1.0 µg/kg (N=4) | Part A: Romiplostim 3 µg/kg (N=4) | Part A: Romiplostim 6 µg/kg (N=4) | Part A: Romiplostim 10 µg/kg (N=4) | Part B: Placebo (N=4) | Part B: Romiplostim 1.0 µg/kg (N=8) | Part B: Romiplostim 3.0 µg/kg (N=8) | Part B: Romiplostim 6.0 µg/kg (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 4 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Loose stools (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 1
Oral mucosal petechiae (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0
Tongue haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Fibrosis (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Venipuncture site bruise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 3 | 3 | 3 | 2 | 6 | 3 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 2 | 3 | 4 | 1 | 0 | 0 | 2 | 3 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ejaculation disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Premenstrual syndrome (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 3 | 4 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 2 | 3 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash scaly (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Petechiae (Vascular disorders) | 0 | 2 | 1 | 2 | 2 | 1 | 1 | 3 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vascular insufficiency (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.